CLINICAL TRIAL: NCT03100240
Title: The Preliminary Mechanism Study of Modified Utral-long Protocol in Improving Endometrial Receptivity in Patients With PCOS and Insulin Resistance
Brief Title: The Mechanism of Modified Utral-long Protocol in Improving Endometrial Receptivity in Patients With PCOS and IR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: It is difficult to recruit patients.
Sponsor: Reproductive & Genetic Hospital of CITIC-Xiangya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 81501328
Record Dates: First submitted 2017-03-20; First posted 2017-04-04 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: PCOS

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental group (Experimental): Modified Supper Long Protocol
  Interventions: Procedure: Modified Supper Long Protocol
- control group (No Intervention): long protocol

INTERVENTIONS:
Procedure: Modified Supper Long Protocol — In Modified Supper Long Protocol, GnRH-a was used twice in mid-luteal phaes
  Arms: Experimental group

SUMMARY:
NF-κB pathway activation-induced endometrial insulin resistance was one of the causes of infertility patients with PCOS and insulin resistance whose endometrial receptivity is declined .The investigators' previous findings indicated that the use of modified utral-long protocols ( GnRH-a was used twice in mid-luteal phaes) can improve clinical outcomes by improving endometrial receptivity in patients with PCOS , but the mechanism was not clear. Previous research also found that GnRH-a reduced the activity of NF-κB pathway in endometrial stromal cells and depended the dose and time.Thus, The investigators' subject will try to applicate GnRH-a to explore the influence of NF-κB pathway activity 、the state of insulin resistance and embryo implantation rate ;then we will investgate GnRH-a whether reduce NF-κB pathway activity-induced insulin resistance and ultimately improve endometrial receptivity by using GnRH-a in infertility patients with PCOS and insulin resistance.The investigators' research attempt to provide ideas for seeking inflammatory medication target in assisted reproductive technology in patients with PCOS by exploring the immune mechanism of GnRHa on improving the endometrial receptivity .

DETAILED DESCRIPTION:
The endometrial biopsy was performed in the previous cycle of the protocol. According to the expression of NF-κB in the endometrium random group. The difference of NF - κB expression in patients with different protocol were compared.

ELIGIBILITY:
Inclusion Criteria:

* age<36years,
* PCOS,
* Insulin resistance (HOMA-IR = fasting insulin (FINS) × fasting blood glucose (FPG) / 22.5, HOMA-IR ≥ 2.69 ）;

Exclusion Criteria:

* uterine abnormalities (double uterus, bicornuate uterus, unicornuate uterus and uterine mediastinum),
* intrauterine adhesions,
* endometriosis, adenomyosis,
* Hydrosalpinx,
* uterine fibroids (submucosal fibroids, non-mucosal fibroids > 4 cm and / or endometrial pressure),
* Hyroid dysfunction and hyperprolactinemia.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate | 28 days after transplantation
  a beating heart tube was 99 detected by ultrasound examination

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive & Genetic Hospital of CITIC-XIANGYA, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided